CLINICAL TRIAL: NCT06075199
Title: A Prospective Cohort Study for Gastric Cancer Prediction in Patients With Intestinal Metaplasia
Brief Title: Intestinal Metaplasia Cohort for Gastric Cancer Prediction
Status: Recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Soo-Jeong Cho, Professor, Seoul National University Hospital
Other Study IDs: 2307-061-1448
Record Dates: First submitted 2023-10-03; First posted 2023-10-10 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Intestinal Metaplasia of Gastric Mucosa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Gastric mucosal tissue from the antrum and body of the stomach
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study, we aim to establish a prospective cohort of patients with endoscopically and histologically confirmed intestinal metaplasia, collect gastric mucosal tissue samples from this cohort, and follow the development of gastric cancer over time.

DETAILED DESCRIPTION:
Patients visiting Seoul National University Hospital, who have previously received an incidental diagnosis of intestinal metaplasia during a prior gastroscopy examination, will be considered as potential candidates for this study. Upon obtaining their informed consent to participate, the initial endoscopy procedure will involve the collection of biopsies to ensure an accurate histological diagnosis of intestinal metaplasia. These biopsies will be taken from the antrum and body of the stomach, according to the protocol of the updated Sydney system, to pathologically diagnose the extent and severity of intestinal metaplasia. One to two pieces of tissue remaining from this diagnostic process will be retained for future analysis. Subsequently, patients will be followed up on an outpatient basis to track the development of gastric cancer through routine screening endoscopies. In cases where patients develop gastric cancer, a comparative analysis will be conducted with those who do not develop gastric cancer, to determine the differences in expression of markers in the gastric mucosal tissue that was collected during the initial endoscopy. Our ultimate aim is to identify potential biomarkers that may serve as predictive indicators for the development of gastric cancer in patients with a preexisting diagnosis of intestinal metaplasia.

ELIGIBILITY:
Inclusion Criteria:

* Patients who visit Seoul National University Hospital
* Patients who have been visually diagnosed with intestinal metaplasia at a prior exam

Exclusion Criteria:

* Patients who have been previously diagnosed with gastric cancer or adenoma
* Patients who have previously received gastrectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatient clinic visitors
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-09-13 (Actual); Primary Completion 2033-06-30 (Estimated); Study Completion 2033-06-30 (Estimated)

PRIMARY OUTCOMES:
Gastric Cancer Development | 10 years
  Number of Participants Who Develop Gastric Cancer

CONTACTS AND LOCATIONS:
Overall Officials: Soo-Jeong Cho, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea